CLINICAL TRIAL: NCT06948604
Title: Impact of Kegel Exercises on the Postoperative Outcomes of Patients Undergoing Transurethral Resection of the Prostate
Brief Title: Impact of Kegel Exercise on Patient Outcomes Post TURP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hazem Tarraf Abo Dief, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: kegel exercise and TURP outcom
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-04

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
Keywords: Kegel exercise,TURP, Patient outcomes and BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kegel exercise (Other): kegel exercise improve muscles strength
  Interventions: Behavioral: Exercise
- study group and control group (Experimental): kegel exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — this exercise used to improve urine complication post TURP

SUMMARY:
how kegel exercise will improve patient outcomes by reducing post TURP LUTs , improve patient performance status and improve patient self esteem

DETAILED DESCRIPTION:
patients will divided in to two group study and control, study group will perform kegel exercise postoperative and follow patient progress at 1, 3,6 month while control group receive routine care

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with BPH and undergoing TURP
* Patient age range from 45-65years old
* Patient understand verbal and written instructions

Exclusion Criteria:

Patient confirmed diagnosis with prostate cancer (biopsy-PSA) Conversion to open prostatectomy Patient has cognitive impairment Patient has chronic cough /chronic bronchitis or asthma

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male patient only
Enrollment: 92 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score | within 3 month
  This tool was developed by Barry et al., (1992) for assessing LUTs after TURP. Post-TURP, patients may continue to experience urinary symptoms such as frequency, urgency, nocturia, and incomplete emptying. International Prostate Symptom Score consists of seven symptom-related questions and one quality-of-life question to assess the severity of LUTs. The symptom questions evaluate incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia, each scored from 0 (never),1(less than 1time in 5), 2 (less than half the time), 3 (about half the time), 4 (more than half the time) to 5 (almost always), with a total score ranging from 0 to 35 (mild: 0-7, moderate: 8-19, severe: 20-35).

SECONDARY OUTCOMES:
World Health Organization Performance Status Scale | within 6 month
  It developed by Oken et al., (1982) to assess how disease affects daily living abilities of patient and describes the status of symptoms and functions. It consists of: Grade 0: Normal activity, Grade 1: Restricted in physical strenuous activities but ambulatory and able to carry out work of light or sedentary nature, Grade 2: Less than 50% of daytime in bed, Grade 3: More than 50% of daytime in bed, Grade 4: Completely disabled and Grade 5: Dead.

IPD SHARING:
Plan to Share IPD: Undecided